CLINICAL TRIAL: NCT02817893
Title: Comparison of Respiratory Variations of the Pulse Oximetry Plethysmographic Raw Signal and Pulse Pressure During Abdominal Surgery (PLETHYSMO)
Acronym: PLETHYSMO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D22215
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Abdominal Surgery
Keywords: ∆POP: variation of the plethysmographic waveform of pulse oximetry; ∆PP: pulse pressure variation; pulse oximetry plethysmographic; abdominal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The waveform plethysmographic signal can be used to establish an index for predicting fluid responsiveness (∆POP: respiratory variation of the plethysmographic waveform of pulse oximetry). This index was validated in some studies and because of its non-invasiveness it seems very interesting in anesthesia.

However, in a previous study the investigators evaluated the correlation between the results provided by this index (∆POP) and those of the reference index (∆PP: pulse pressure variation), and the obtained results were significantly lower than what had been previously described. In this study, the index was calculated from a recording of a filtered signal. This unavoidable application of a filter on anesthesia monitors could contribute to the discrepancy between the ∆POP and the ∆PP.

The realization of a new study, comparing ∆PP and ∆POP obtained from an unfiltered plethysmographic signal, should answer the ∆POP ability to be used in place of ∆PP.

ELIGIBILITY:
Inclusion Criteria:

* Hospital patient in general surgery and digestive department
* Adult
* Digestive sus mesocolic surgery with direct abdominal approach justifying a semi-invasive hemodynamic monitoring by arterial catheterization (liver, pancreatic, gastric and duodenal surgery)
* Surgical approach by laparotomy
* Patient under general anesthesia with mechanical ventilation
* Agreeing to participate in the study after receiving information note

Exclusion Criteria:

* Known left systolic ventricular and/or diastolic failure
* Arrhythmias
* Surgery performed with thoracic approach
* Surgery by laparoscopy
* Emergency surgery
* Hypersensitivity or allergic to any of the product used for usual anesthesia, hypersensitivity to soya or egg lecithin
* Personal or familial history of malignant hyperthermia
* Severe kidney impairment (creatinin clearance <30ml/min)
* Patients who participated in the previous month to another study protocol
* Pregnant women or nursing
* Under-age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo sus mesocolic surgery under general anesthesia and by direct approach, whose anesthesic management requires continuous monitoring of blood pressure (arterial catheter).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
∆PP: pulse pressure variation | Day 0
  reference index measured during abdominal surgery
∆POP: respiratory variation of the plethysmographic waveform of pulse oximetry | Day 0
  noninvasive index obtained from plethysmographic raw signal measured during abdominal surgery